CLINICAL TRIAL: NCT06726330
Title: Evaluation of Risk Control of Advanced Stage Tubo-ovarian or Primary Peritoneal Carcinoma Associated With Ovarian Carcinoma Risk-reducing Strategies, Including Fimbriectomy With Delayed Oophorectomy, in Women With a Germline Mutation Predisposing to Ovarian or Pelvic Cancer
Brief Title: Risk-reducing Strategies, Including Fimbriectomy, in Women With a Germline Mutation Predisposing to Ovarian or Pelvic Cancer
Acronym: FIMBRIMENOP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FIMBRIMENOP-2402; PHRC-K24-013 (Other Grant/Funding Number: INca); 2024-A01760-47 (Other: ANSM)
Record Dates: First submitted 2024-11-25; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Tubo-ovarian Carcinoma; High-grade Serous Carcinoma; Primary Peritoneal Carcinoma Stage III; Primary Peritoneal Carcinoma Stage IV; Primary Peritoneal Carcinoma
Keywords: Tubo-ovarian carcinoma; Primary peritoneal carcinoma; BRCA1/2 mutations; RAD51C/D mutations; PALB2 mutation; Preventive surgery; Fimbriectomy; Bilateral salpingo-oophorectomy; BSO; Cancer prevention; Premenopausal women; Genetic predisposition to cancer
MeSH Terms: interventions — Sterilization, Tubal

STUDY DESIGN:
Intervention Model Description: This is a non-randomized controlled preference trial. Participants decide their surgical approach based on counseling. The study accommodates real-world clinical practices, empowering patients in the decision-making process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fimbriectomy Followed by Delayed Oophorectomy (F-DO) (Experimental): Participants in this arm will undergo fimbriectomy, a surgical procedure to remove the fimbrial end of the fallopian tubes, while preserving ovarian function. A delayed oophorectomy (removal of the ovaries) will be performed at menopause or later, based on individual timing and preferences. This approach aims to reduce the risk of advanced-stage tubo-ovarian or primary peritoneal carcinoma while minimizing the adverse effects of premature menopause.
  Interventions: Procedure: Fimbriectomy Followed by Delayed Oophorectomy (F-DO)
- Bilateral Salpingo-Oophorectomy (BSO) (Active Comparator): Participants in this arm will undergo a bilateral salpingo-oophorectomy (BSO), the standard preventive surgical strategy, involving the removal of both fallopian tubes and ovaries. This procedure is performed around the recommended age of 40-45 years for women with BRCA1/2 mutations or similar high-risk genetic predispositions. The primary objective is to eliminate the risk of tubo-ovarian or primary peritoneal carcinoma, though it induces premature menopause.
  Interventions: Procedure: Bilateral Salpingo-Oophorectomy

INTERVENTIONS:
Procedure: Fimbriectomy Followed by Delayed Oophorectomy (F-DO) — This intervention involves two stages:
  1. Fimbriectomy: A preventive surgical procedure that removes the fimbrial end of the fallopian tubes, including adjacent ovarian tissue, while preserving ovarian function to avoid premature menopause.
  2. Delayed Oophorectomy: The removal of ovaries, performed at menopause or later, depending on patient preference and clinical guidelines.
     * The F-DO strategy aims to reduce the risk of tubo-ovarian or primary peritoneal carcinoma, which often originates in the fallopian tubes, while minimizing the adverse effects of premature menopause such as cardiovascular disease and osteoporosis
  Other Names: fimbriectomy
  Arms: Fimbriectomy Followed by Delayed Oophorectomy (F-DO)
Procedure: Bilateral Salpingo-Oophorectomy — This standard surgical intervention involves the removal of both fallopian tubes and ovaries (BSO) to eliminate the risk of tubo-ovarian or primary peritoneal carcinoma. It is typically recommended for women with a genetic predisposition (e.g., BRCA1/2 mutations) around the age of 40-45. While highly effective in preventing cancer, BSO induces premature menopause, which may result in long-term side effects such as increased cardiovascular risk, osteoporosis, and cognitive decline.
  Other Names: BSO
  Arms: Bilateral Salpingo-Oophorectomy (BSO)

SUMMARY:
• FIMBRIMENOP-2402 study aims to evaluate the long-term management of cancer risks in premenopausal women who have a genetic predisposition to tubo-ovarian or primary peritoneal carcinoma, such as mutations in BRCA1, BRCA2, RAD51C, RAD51D, or PALB2 genes. This study offers an alternative to standard preventive surgery (bilateral salpingo-oophorectomy or BSO) by exploring the use of fimbriectomy (removal of the fallopian tube's fimbria) followed by delayed oophorectomy (removal of ovaries at menopause).

It's a pragmatic multicenter trial conducted across various medical centers, employing a non-randomized controlled preference design to compare two preventive surgical strategies:

1. Fimbriectomy followed by delayed oophorectomy (F-DO).
2. Bilateral salpingo-oophorectomy (BSO).

The primary objective is to compare the long-term efficacy of two preventive surgical strategies :

1. Fimbriectomy followed by delayed oophorectomy (F-DO).
2. Bilateral salpingo-oophorectomy (BSO).

As for the design of the study, participants choose their preferred surgical strategy during or after oncogenetic counseling, ensuring patient autonomy in decision-making.

• Follow-Up: Long-term follow-up includes clinical assessments, data collection from medical networks, and integration with national health databases to track outcomes up to the age of 70.

This is the first French comparative study in real-world settings and is classified as interventional research (RIPH1) under French regulations, given the need to validate fimbriectomy efficacy.

DETAILED DESCRIPTION:
* The FIMBRIMENOP-2402 study is a pragmatic, multicenter, interventional trial (RIPH1) designed to evaluate long-term management strategies for reducing cancer risk in premenopausal women genetically predisposed to tubo-ovarian or primary peritoneal carcinoma. Women carrying mutations in BRCA1, BRCA2, RAD51C, RAD51D, or PALB2 genes are the primary focus of this investigation.
* Objectives

The primary objective is to evaluate, on a long-term horizon, the control of the risk of advanced stage tubo-ovarian or primary peritoneal carcinoma according to the chosen care pathway, and more specifically whether F-DO is non inferior to BSO, in women with a germline mutation predisposing to the risk of high grade serous tubo-ovarian or primary peritoneal carcinoma.

The study aims to determine whether F-DO is non-inferior to BSO in controlling the risk of advanced-stage tubo-ovarian or primary peritoneal carcinoma in high-risk women.

The secondary objectives include evaluating the benefit-risk ratio of these approaches by assessing:

* Menopause-related side effects, such as cardiovascular and osteoporosis-related events.
* Surgical complications and overall survival.
* Long-term oncological outcomes, including breast cancer risks.
* Patient-reported preferences and compliance with the chosen pathway.

The study will also contribute to a prospective meta-analysis of similar international studies.

• Design and Methodology

The study employs a non-randomized controlled preference design, allowing participants to choose their preventive surgical strategy after informed counseling with oncogeneticists and gynecologic surgeons. This approach promotes patient autonomy while reflecting real-world clinical decision-making. Participants may revise their choice at any time before the first surgical intervention. The actual treatment received or the final preference will define the "care pathway".

• Population and Recruitment

The study will enroll 1,100 premenopausal women aged 35-50 years from multiple French centers, all of whom are at an elevated genetic risk for tubo-ovarian or primary peritoneal carcinoma. Recruitment is expected to span five years, with follow-up continuing until participants reach 70 years of age.

• Data Collection and Follow-Up

Data collection integrates multiple sources to ensure comprehensive coverage of outcomes:

1. Annual Clinical Assessments: Participants undergo routine clinical evaluations, including physician visits, medical reports, and online questionnaires or phone interviews.
2. Regional Oncogenetic Networks: Data from regional networks are incorporated to monitor oncological events and compliance.
3. French Administrative Health Database (SNDS): Extraction of anonymized health records ensures the completeness of reported events and reduces logistical complexity.

   * Endpoints :
   * Primary Endpoint :

The incidence of advanced-stage (stage III or IV) tubo-ovarian or primary peritoneal carcinoma, measured as the time from study entry to the occurrence of cancer, with death without cancer as a competing event. Censoring will occur at the last follow-up visit for women without cancer.

* Secondary Endpoints include :
* Incidence of tubo-ovarian carcinoma at any stage, breast cancer, cardiovascular and osteoporosis-related events.
* Age at menopause.
* Surgical complications within 30 days post-surgery, graded per NCI-CTCAE V5.0.
* Statistical Analysis

The final analysis will occur when all participants have been followed for 35 years, with interim analyses planned every six years or upon reporting of 10 events. Data will be analyzed to compare oncological outcomes, quality of life, and survival between the F-DO and BSO groups. Biases inherent in the preference design will be addressed through appropriate statistical modeling.

• Ethical Considerations

The study adheres to French regulatory requirements, including patient data confidentiality under the GDPR and ethical review by relevant committees. Informed consent will be obtained from all participants, with clear communication of risks and benefits.

By evaluating the efficacy and safety of F-DO, this study has the potential to redefine preventive surgical strategies, optimizing outcomes for women at high genetic risk of ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Woman between 35 to 50 years
2. Addressed to or followed in an oncogenetic counselling
3. Identified risk of tubo-ovarian or primary peritoneal carcinoma based on mutational status (BRCA1, BRCA 2, RAD51C, RAD51D, PALB2). The list of considered mutations may be extended during the study.
4. Written informed consent
5. Patient covered by the French "Social Security"

Exclusion Criteria:

1. Prior bilateral oophorectomy and/or bilateral salpingectomy for any reason (prophylactic surgery or other)
2. Personal history of ovarian, fallopian tube or primary peritoneal cancer
3. Menopause defined by

   • In women without prior chemotherapy If no prior hysterectomy: the absence of menses for at least 12 months, or FSH > 20 UI/L with low estrogen level with no identified gynecological or endocrine explanation. Amenorrhea related to an intrauterine device, vaginal ring or estrogen-progestin pill will not be considered as menopause.

   If prior hysterectomy: FSH >20 UI/L with low estrogen level (with or without vasomotor symptoms, genitourinary symptoms)
   * In women with prior chemotherapy: the absence of menses for at least 24 months
   * In all women with progesterone-loaded intra-uterine device (IUD): FSH > 20 UI/L with low estrogen level
4. Inability to comply with medical follow-up of the trial (geographical, social or psychological reasons)
5. Patient under guardianship or curatorship

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1100 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2065-03 (Estimated); Study Completion 2065-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Advanced-Stage (Stage III or IV) Tubo-Ovarian or Primary Peritoneal Carcinoma | Up to 70 years of age
  The study evaluates the long-term incidence of advanced-stage (Stage III or IV) tubo-ovarian or primary peritoneal carcinoma. This measure will be assessed using annual clinical evaluations, patient questionnaires, medical records, and data extracted from the French National Health Database (SNDS) and regional oncogenetic networks. Time from study entry to cancer diagnosis will be calculated, with death without cancer considered as a competing event. Data will be censored at the last follow-up visit for participants alive without cancer.

SECONDARY OUTCOMES:
Incidence of Any-Stage Tubo-Ovarian or Primary Peritoneal Carcinoma | Up to 70 years of age
  Time from study entry to diagnosis of any stage of tubo-ovarian or primary peritoneal carcinoma, including pre-invasive lesions such as serous tubal intraepithelial carcinoma (STIC).
Age at Menopause | Over the study period (up to age 70).
  The age at menopause will be determined through clinical assessments, hormone level measurements, and patient-reported outcomes. Criteria include cessation of menses for at least 12 months in non-hysterectomized women or FSH levels >20 UI/L with low estrogen levels.
Incidence of Cardiovascular Events and Osteoporosis-Related Events | Over the study period (up to age 70)
  Long-term cardiovascular (e.g., myocardial infarction, stroke) and osteoporosis-related events (e.g., hip fractures) will be recorded from clinical evaluations and the SNDS database.
Overall Survival | From study entry to death from any cause.
  Overall survival will be tracked using clinical data, SNDS records, and vital status updates.
Surgical Complications | 30 days following the surgery
  Complications will be graded using the NCI-CTCAE v5.0 system and classified as related to surgery. Severe adverse events (grade 3+) and serious adverse events will be reported.

OTHER OUTCOMES:
Benefit-Risk Ratio Analysis | Over the study period (up to age 70)
  Composite analysis of event-free survival, including advanced-stage tubo-ovarian or primary peritoneal carcinoma, breast cancer, cardiovascular events, osteoporosis-related events, and death from any cause. This measure integrates the oncological and quality-of-life impacts of the surgical strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos MARTINEZ GOMEZ, MD, Study Director — Centre Oscar Lambret; Audrey MAILLIEZ, MD, Study Director — Centre Oscar Lambret
Locations (23):
- France (23):
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Universitaire Dijon Bourgogne, Dijon
  - Centre hospitalier universitaire Grenoble-Alpes, Grenoble
  - Centre Hospitalier Universitaire de Lille, Lille
  - Centre Oscar Lambret, Lille
  - Clinique du Bois, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Institut de cancérologie de l'Ouest Centre René GAUDUCHEAU, Nantes
  - Centre Antoine Lacassagne, Nice
  - Gustave Roussy, Paris
  - Hôpital de la Pitié Salpêtrière - AP-HP, Paris
  - Hôpital Institut CURIE, Paris
  - Hôpital Tenon AP-HP, Paris
  - Institut Godinot, Reims
  - Centre Henri Becquerel, Rouen
  - Hôpitaux Privés Rouennais, Rouen
  - Hôpital de Saint-Cloud, Saint-Cloud
  - Institut universitaire du cancer de Toulouse, Toulouse
  - Hôpital Simone Veil - CH de Troyes, Troyes
  - Centre Hospitalier de Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: Undecided